CLINICAL TRIAL: NCT03820349
Title: Effects of Cystic Fibrosis and Cystic Fibrosis Related Diabetes on Brain Structure and Cognitive Function
Brief Title: Cystic Fibrosis and Cognitive Function
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MED-2018-26438
Record Dates: First submitted 2018-02-26; First posted 2019-01-29 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis
Keywords: CFRD; Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: Subjects with cystic fibrosis
- controls: matched healthy controls

SUMMARY:
The long-term goal of this project is to examine the effects of cystic fibrosis (CF) and cystic fibrosis related diabetes (CFRD) on brain structure and function

DETAILED DESCRIPTION:
A growing body of evidence suggests that hyperglycemia in type 1 and type 2 diabetes is associated with alterations in brain structure and cognitive impairment. People with cystic fibrosis related diabetes (CRFD) are exposed to hyperglycemia as seen in other forms of diabetes, and cystic fibrosis is also associated with chronic systemic inflammation. Both hyperglycemia and chronic inflammation have been postulated to affect brain structure and function. Cystic fibrosis trans-membrane conductance regulator (CFTR). protein is widely expressed in the neurons of the brain including in the hippocampus The hippocampus plays an essential role in learning and memory processing and is thought to be particularly vulnerable to effects of metabolic stressors. The expression of CFTR in neurons has several potential implications for central nervous system function, including cognition.

The long-term goal of this project is to examine the effects of cystic fibrosis (CF) and cystic fibrosis related diabetes (CFRD) on brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

patients with Cystic fibrosis

Exclusion Criteria:

* History of stroke
* History of epilepsy
* History of neurosurgical procedures
* Past or current history of severe psychiatric illness
* Pass or current history of alcohol or substance abuse
* Presence of metallic substances in body or inability to remove before imaging procedure
* History of claustrophobia or known inability to tolerate MRI
* Current pregnancy
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cystic Fibrosis
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
MRI outcome | baseline
  Measure the differences in the microstructure (fractional anisotropy) of hippocampus, comparing subjects with cystic fibrosis and healthy controls

SECONDARY OUTCOMES:
Cognitive function | baseline
  Compare performance on neurocognitive function testing in subjects with cystic fibrosis and healthy controls. Multiple cognitive domains will be examined including intellectual function, processing speed. attention and memory.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Science Institute and Center for Magnetic Resonance Research, University of Minnesota, Minneapolis, Minnesota, United States